CLINICAL TRIAL: NCT00004265
Title: Phase II Study of Weekly Paclitaxel as Second-Line Therapy in Patients With Non-Small Cell Lung Cancer
Brief Title: Paclitaxel in Treating Patients With Recurrent or Refractory Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067524; WCCC-CO-98501; NCI-G00-1669
Record Dates: First submitted 2000-01-28; First posted 2004-07-26 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have recurrent or refractory non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and response duration in patients with recurrent or refractory non-small cell lung cancer (NSCLC) treated with second line paclitaxel. II. Determine the qualitative and quantitative toxicities of this treatment regimen in relapsed patients with recurrent NSCLC. III. Evaluate the time to treatment failure and overall survival in this patient population.

OUTLINE: Patients receive paclitaxel IV over 1 hour weekly for 6 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 30-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non-small cell lung cancer with documented recurrent or refractory disease Progressive disease at more than 3 months from completion of first line chemotherapy OR Progressive disease during first line chemotherapy Clinically stable CNS metastases allowed

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL AST no greater than 5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No clinically significant bradyarrhythmias Other: Neuropathy less than grade 2 Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: See Disease Characteristics Must have had at least 1 prior first line chemotherapy regimen for metastatic or locally advanced disease One prior paclitaxel regimen (every 3 week schedule) allowed if no progressive disease at less than 3 months from completion of therapy At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy (indicator lesions within the radiation port must have progressed since completion of therapy) Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States